CLINICAL TRIAL: NCT01747577
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, and Phase IV Study of Efficacy and Safety of Solifenacin Succinate in Patients With Overactive Bladder After TURP or PVP
Brief Title: Post Marketing Study to Evaluate the Efficacy and Safety of Solifenacin in Patients With OAB (Overactive Bladder) After TURP (Trans-urethral Resection of Prostate) or PVP (Photoselective Vaporization of Prostate)
Acronym: POST-TURP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VC-OAB-12-01
Record Dates: First submitted 2012-12-10; First posted 2012-12-11 (Estimated); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Overactive Bladder; Benign Prostate Hyperplasia; Transurethral Resection of Prostate; Photoselective Vaporization Prostatectomy
Keywords: Muscarine antagonist; Prostatectomy; Uroflowmetry
MeSH Terms: conditions — Urinary Bladder, Overactive; Prostatic Hyperplasia | interventions — Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Solifenacin group (Experimental)
  Interventions: Drug: Solifenacin Succinate
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Solifenacin Succinate — Oral
  Other Names: YM905; Vesicare®
  Arms: Solifenacin group
Drug: Placebo — Oral
  Arms: Placebo group

SUMMARY:
The purpose of this study is to demonstrate superiority of the solifenacin succinate (treatment) over the placebo (control) based on the change from the baseline in the mean number of urgency episodes per 24 hours after 2 weeks.

DETAILED DESCRIPTION:
The BPH (benign prostate hyperplasia) patients who have OAB (overactive bladder) after TURP (trans-urethral resection of prostate) or PVP (photoselective vaporization of prostate) will participate in this study. The subjects will be randomized 1:1 to the solifenacin succinate group or to the placebo treatment group. The subjects shall take investigational product each night before sleeping from for four weeks and complete voiding diary. At Week-2 and Week-4 of the treatment, the subjects will be asked to complete the following activities: physical exam, vital signs test, IPSS, OABSS, post-void residual (PVR) test, and uroflowmetry, and will be asked to answer the BSW, (Benefit, Satisfaction and Willingness to Continue Questions) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Screening

  * Patients who are willing and able to accurately complete the voiding diary, IPSS, and OABSS
  * Patients who have been diagnosed with BPH and are scheduled to receive TURP or PVP
* Randomization (after TURP or PVP)

  * Patients who have been diagnosed with OAB by the investigators
  * Patients who underwent catheter removal 5±2 days beforehand and will have more than an average of three urgency episodes per 24 hrs and more than an average of eight micturitions per 24 hrs in a row before Visit 3, as recorded in the voiding diary
  * Patients who will score more than 5 in questions 2, 4, and 7, which are on the storage symptoms in IPSS
  * Patients who will score more than 4 in question 3 and more than 5 in the OABSS
  * Patients who have not been treated with any medication for overactive bladder (OAB) symptoms 14 days before the randomization

Exclusion Criteria:

* Screening

  * Patients who have been diagnosed with prostate cancer or bladder cancer and who have a present or resolved malignant disease in any pelvic organ
  * Patients who have neurological diseases that affect micturition and can cause neurogenic bladder disease such as multiple sclerosis, Parkinson's disease, severe cerebral arteriosclerosis, dementia, stroke, or myelitis
  * Patients who have had serious adverse events or are hypersensitive to anticholinergics
  * Patients who have a severe gastrointestinal obstruction disease such as toxin megacolon, ulcerative colitis, intestinal atonia, paralytic ileus, and gastric retention
  * Patients who have been diagnosed with severe myasthenia
  * Patients who have been diagnosed with narrow-angle glaucoma
  * Patients who have serious hepatic impairment (child class C)
  * Patients who are being treated with a CYP3A4 inhibitor (e.g., Ketoconazole)
  * Patients who have severe renal impairment or who are undergoing hemodialysis
  * Patients who have diabetic neuropathy
  * Patients who have a significant urinogenital disease such as UTI, interstitial cystitis, urothelial tumor, bladder stone, or urinary retention
  * Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
  * Patients who have another medical or psychiatric condition that will make them inappropriate for participate in this study in the opinion of the investigators
  * Patients who have participated in other clinical trials within 30 days before the screening visit
* Randomization

  * Patients who have been diagnosed with clinically significant bladder outlet obstruction by investigators
  * Patients whose PVR is greater than 100 mL
  * Patients who have been diagnosed with prostate cancer or bladder cancer and who have a present or resolved malignant disease in any pelvic organ
  * Patients who have neurological diseases that affect micturition and can cause neurogenic bladder disease such as multiple sclerosis, Parkinson's disease, severe cerebral arteriosclerosis, dementia, stroke, or myelitis
  * Patients who have had serious adverse events or are hypersensitive to anticholinergics
  * Patients who have a severe gastrointestinal obstruction disease such as toxin megacolon, ulcerative colitis, intestinal atonia, paralytic ileus, and gastric retention
  * Patients who have been diagnosed with severe myasthenia
  * Patients who have been diagnosed with narrow-angle glaucoma
  * Patients who have serious hepatic impairment (child class C)
  * Patients who are being treated with a CYP3A4 inhibitor (e.g., Ketoconazole)
  * Patients who have severe renal impairment or who are undergoing hemodialysis
  * Patients who experienced severe side effects after their operation
  * Patients who have diabetic neuropathy
  * Patients who have a significant urinogenital disease such as UTI, interstitial cystitis, urothelial tumor, bladder stone, or urinary retention
  * Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
  * Patients who have another medical or psychiatric condition that will make them inappropriate for participate in this study in the opinion of the investigators
  * Patients who have participated in other clinical trials within 30 days before the screening visit

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-12-04 (Actual); Primary Completion 2013-10-24 (Actual); Study Completion 2013-10-24 (Actual)

PRIMARY OUTCOMES:
Mean change from the baseline in the number of urgency episodes per 24 hrs in the voiding diary at Week 2 | Baseline and at week 2

SECONDARY OUTCOMES:
Mean change from the baseline in the number of urgency episodes per 24 hrs in the voiding diary at Week 4 | Baseline and at week 4
Change from baseline in IPSS total score | Baseline, at week 2 and at week 4
  IPSS: International Prostate Symptom Score
Changes from baseline in IPSS storage subscale score | Baseline, at week 2 and at week 4
Changes from baseline in IPSS voiding subscale score | Baseline, at week 2 and at week 4
Changes from baseline in individual IPSS scores | Baseline, at week 2 and at week 4
Changes from baseline in IPSS QOL | Baseline, at week 2 and at week 4
  QOL: Quality of Life
Changes from baseline in OABSS total score | Baseline, at week 2 and at week 4
  OABSS: OverActive Bladder Sympton Score
Change from baseline in average number of micturitions per 24 hrs for three days as recorded in the voiding diary | Baseline, at week 2 and at week 4
Safety assessed by the incidence of adverse events, physical exam, and vital signs | For 4 weeks of the treatment
Urinal post voiding residual volume | Before treatment at week 2 and at week 4
  Measured by ultrasound or bladder scan
Maximum flow rate of the urine | Before treatment at week 2 and at week 4
  Assessment using uroflowmetry

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results Web site — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=VC-OAB-12-01